CLINICAL TRIAL: NCT05892497
Title: Effectiveness of Tecarterapy on the Performance of Amateur Athletes
Brief Title: Tecarterapy on the Performance of Amateur Athletes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxim Canet Vintró (Other)
Responsible Party: Sponsor-Investigator, Maxim Canet Vintró, Principal investigator, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBAS-2021-08
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Diathermy Plate Burn; Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tecartherpay Group (Experimental): A single 25-minute tecartherapy procedure will be performed in both legs with the T-Plus Wintecare® machine. The configuration of the tecartherapy programme will be in 40 watts resistive mode for each muscle.
  Interventions: Other: Tecartherapy
- Sham group (Sham Comparator): The same procedure of the intervention group will be performed but with the tecartherapy machine without power (sham). The machine will be on but no power will be supplied.
  Interventions: Other: Tecartherapy

INTERVENTIONS:
Other: Tecartherapy — The tecartherapy intervention was with a deep diathermy machine applied to the patient's lower extremity for 30 minutes.

SUMMARY:
Physical therapies based on electrical or electromagnetic stimulation have been used in rehabilitation, in some cases combining electrical therapy with radiofrequency. Specifically, resistive capacitive electrical transfer therapy (CRet) has been used in physical rehabilitation and sports medicine to treat muscle, bone, ligament and tendon injuries. CRet is a non-invasive electrothermal therapy classified as deep thermotherapy, which is based on the application of electrical currents within the radiofrequency range of 300 kHz - 1.2 MHz. While the heat conducted by surface thermotherapy cannot reach the muscle due to the electrical resistance of the tissues, the capacitive-resistive electrical currents in CRet therapy can generate heating of deep muscle tissues, which in turn improves haemoglobin saturation. In Europe, CRet is widely used in various medical rehabilitation processes. The physiological effects of this type of physiotherapy are generated by the application of an electromagnetic field with a frequency of approximately 0.5 MHz to the human body. The effects attributed to this technique include increased deep and superficial blood circulation, vasodilatation, increased temperature, removal of excess fluid and increased cell proliferation.

Some of these reactions, such as increased blood perfusion, are known to be related to the increase in temperature, but others, such as increased cell proliferation, appear to be primarily related to the passage of current.

It is also true that this increase in tissue temperature, generated through the application of the device, is a physical reaction to the passage of current (Joule effect). Although there is already clinical literature supporting this mechanism, the amount of energy and current that must be transferred to obtain the desired temperature rise is unknown. Moreover, the control of these reactions, by adjusting parameters such as absorbed power and electrode position, is still largely based on the empirical experience of therapists .

Recently, new cadaveric publications have been generated, which support the mechanisms of current flow and thermal changes in this situation.

Against this background, in which thermal effects, current passage and symptomatic improvements have been demonstrated in patients with pathology, the possibility that these treatments may improve functional sporting abilities is raised. This hypothesis arises from the fact that current flow and thermal changes have been directly related to viscoelastic changes in capsular and muscle tissue.

To date, there is no study that has assessed whether this therapy generates any change in functional variables related to sports performance in professional athletes.

DETAILED DESCRIPTION:
Physical therapies based on electrical or electromagnetic stimulation have been used in rehabilitation, in some cases combining electrical therapy with radiofrequency. Specifically, resistive capacitive electrical transfer therapy (CRet) has been used in physical rehabilitation and sports medicine to treat muscle, bone, ligament and tendon injuries. CRet is a non-invasive electrothermal therapy classified as deep thermotherapy, which is based on the application of electrical currents within the radiofrequency range of 300 kHz - 1.2 MHz. While the heat conducted by surface thermotherapy cannot reach the muscle due to the electrical resistance of the tissues, the capacitive-resistive electrical currents in CRet therapy can generate heating of deep muscle tissues, which in turn improves haemoglobin saturation. In Europe, CRet is widely used in various medical rehabilitation processes. The physiological effects of this type of physiotherapy are generated by the application of an electromagnetic field with a frequency of approximately 0.5 MHz to the human body. The effects attributed to this technique include increased deep and superficial blood circulation, vasodilatation, increased temperature, removal of excess fluid and increased cell proliferation.

Some of these reactions, such as increased blood perfusion, are known to be related to the increase in temperature, but others, such as increased cell proliferation, appear to be primarily related to the passage of current.

It is also true that this increase in tissue temperature, generated through the application of the device, is a physical reaction to the passage of current (Joule effect). Although there is already clinical literature supporting this mechanism, the amount of energy and current that must be transferred to obtain the desired temperature rise is unknown. Moreover, the control of these reactions, by adjusting parameters such as absorbed power and electrode position, is still largely based on the empirical experience of therapists .

Recently, new cadaveric publications have been generated, which support the mechanisms of current flow and thermal changes in this situation.

Against this background, in which thermal effects, current passage and symptomatic improvements have been demonstrated in patients with pathology, the possibility that these treatments may improve functional sporting abilities is raised. This hypothesis arises from the fact that current flow and thermal changes have been directly related to viscoelastic changes in capsular and muscle tissue.

To date, there is no study that has assessed whether this therapy generates any change in functional variables related to sports performance in professional athletes.

ELIGIBILITY:
Inclusion Criteria:

* Athletes between 18 and 30 years of age (athletics and field sports such as soccer, basketball, rugby... that may involve sprinting) federated and competing in university or national amateur leagues that perform sprinting and jumping in their sports practice.
* Active participation in regional, national or international competitions.
* Study participants must have signed the informed consent form in order to evaluate their inclusion in the study.

Exclusion Criteria:

* Volunteers who have suffered a sports injury during the last two months or are unable to perform physical activity.
* Not understanding the information provided by the therapist.
* Participate in other research studies.
* Being under a pharmacological medical treatment that may interfere with the measures, such as treatment with anticonvulsants, antidepressants, etc.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in 30 meters sprint (seconds) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  Photoelectric cells will be used to measure the time required to complete a 30-meter sprint.
Changes in electromyographic activity during sprint (μ/v) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  The mean electromyographic activity of the quadriceps musculature during sprint will be measured with The mDurance® system device (mDurance Solutions SL, Granada, Spain).

SECONDARY OUTCOMES:
Countermovement jump (cm) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  A bipodal jump will be performed and measured with the validated application "MyJump 2"
Changes in electromyographic activity during countermovement jump (μ/v) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  The mean electromyographic activity of the quadriceps musculature during the jump will be measured with The mDurance® system device (mDurance Solutions SL, Granada, Spain).
Changes in isometric leg extension (Newtons) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  A precision dynamometer (Microfeet II) will be used and the maximum force during an isometric contraction of this musculature during 5 seconds of the quadriceps will be analyzed.
Changes in electromyographic activity during isometric leg extension (μ/v) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  The mean electromyographic activity of the quadriceps musculature during the isometric leg extension will be measured with The mDurance® system device (mDurance Solutions SL, Granada, Spain).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain